CLINICAL TRIAL: NCT00388895
Title: Positive Ph Acute Lymphoblastic Leucemia With Intensive Induction Chemotherapy and Glivec, Before and After the Hematopoetic Progenitor Transplant
Brief Title: Glivec in Ph Positive Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BES02; 02-0207 (nº AEMPS)
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Acute Lymphoblastic Leukemia; Cromosome Philadelphia Positive
Keywords: Acute lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Drug Therapy; Imatinib Mesylate

INTERVENTIONS:
Drug: chemotherapy
Drug: Glivec

SUMMARY:
% positive Ph LLA with RC alter the Glivec and induction chemotherapy treatment

DETAILED DESCRIPTION:
Pilot phase II clinical trial, prospective, multicentric and opened

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis LLA Ph+ (BCR/ABL) patients ≤ 65 years old
* Fertile age women must do a pregnancy test in the 7 days previous at the beginning of clinical trial medication
* Performance status 0-2 (Appendix B); Is allowed performance status > 2 because of LLA
* Patients without organ alteration: hepatic function: global bilirubin, AST, ALT, gamma-GT and alkaline phosphatase less than 2 times LSN; renal function: Creatinine < 1,5 mg/dl o Clearance creatinine > 60 ml/min; anormal renal function caused by LLA ; normal heart function (Appendix B): FEV > 50%; No Chronic respiratory illness. If the anormal values are secondary of the experimental illness the investigator can decide himself if the patient can be included at the clinical trial.
* Negative HIV serology
* Written, oral or with witness informed consent. In patients < 18 years old must be signed written and legal representative informed consent.
* No experimental chemotherapy or other experimental treatment. Allowed to begin induction chemotherapy from the diagnosis to confirm Ph. No major surgical process in the previous 14 days of the treatment Start.

Exclusion Criteria:

* Other LLA variability
* Previous history of coronary valvular, hypertensive cardiopathy illness
* Chronic hepatic illness
* Chronic respiratory insufficiency
* Renal insufficiency not caused by LLA
* Severe neurological problems not caused by LLA
* Severe affection of the performance status (grade 3-4 OMS gradation) not caused by LLA
* Pregnancy and women
* Blastic crisis LMC

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2002-06; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
% positive Ph LLA with RC alter the Glivec and induction chemotherapy treatment.
Discover if is possible to treat patients with Glivec plus Standard consolidation treatment.
Discover the Glivec effect over ERM during consolidation treatment and alter transplant

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Chair — Germans Trias i Pujol Hospital
Locations (28):
- Spain (28):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital "Duran I Reynals", Barcelona, Barcelona
  - Hospital "Santa Creu i Sant Pau", Barcelona, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital Universitario "Germans Trias i Pujol", Barcelona, Barcelona
  - Hospital Valle Hebrón-Materno Infantil, Barcelona, Barcelona
  - Hospital Valle Hebrón, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer., Murcia, Murcia
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Carlos Haya, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Oviedo
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Schrappe M, Reiter A, Zimmermann M, Harbott J, Ludwig WD, Henze G, Gadner H, Odenwald E, Riehm H. Long-term results of four consecutive trials in childhood ALL performed by the ALL-BFM study group from 1981 to 1995. Berlin-Frankfurt-Munster. Leukemia. 2000 Dec;14(12):2205-22. doi: 10.1038/sj.leu.2401973. PMID 11187912
- [Background] Thomas X, Thiebaut A, Olteanu N, Danaila C, Charrin C, Archimbaud E, Fiere D. Philadelphia chromosome positive adult acute lymphoblastic leukemia: characteristics, prognostic factors and treatment outcome. Hematol Cell Ther. 1998 Jun;40(3):119-28. PMID 9698220
- [Background] Snyder DS, Nademanee AP, O'Donnell MR, Parker PM, Stein AS, Margolin K, Somlo G, Molina A, Spielberger R, Kashyap A, Fung H, Slovak ML, Dagis A, Negrin RS, Amylon MD, Blume KG, Forman SJ. Long-term follow-up of 23 patients with Philadelphia chromosome-positive acute lymphoblastic leukemia treated with allogeneic bone marrow transplant in first complete remission. Leukemia. 1999 Dec;13(12):2053-8. doi: 10.1038/sj.leu.2401589. PMID 10602428
- [Background] Arico M, Valsecchi MG, Camitta B, Schrappe M, Chessells J, Baruchel A, Gaynon P, Silverman L, Janka-Schaub G, Kamps W, Pui CH, Masera G. Outcome of treatment in children with Philadelphia chromosome-positive acute lymphoblastic leukemia. N Engl J Med. 2000 Apr 6;342(14):998-1006. doi: 10.1056/NEJM200004063421402. PMID 10749961
- [Background] Druker BJ, Tamura S, Buchdunger E, Ohno S, Segal GM, Fanning S, Zimmermann J, Lydon NB. Effects of a selective inhibitor of the Abl tyrosine kinase on the growth of Bcr-Abl positive cells. Nat Med. 1996 May;2(5):561-6. doi: 10.1038/nm0596-561. PMID 8616716
- [Background] Druker BJ, Sawyers CL, Kantarjian H, Resta DJ, Reese SF, Ford JM, Capdeville R, Talpaz M. Activity of a specific inhibitor of the BCR-ABL tyrosine kinase in the blast crisis of chronic myeloid leukemia and acute lymphoblastic leukemia with the Philadelphia chromosome. N Engl J Med. 2001 Apr 5;344(14):1038-42. doi: 10.1056/NEJM200104053441402. PMID 11287973
- [Background] Saffroy R, Lemoine A, Brezillon P, Frenoy N, Delmas B, Goldschmidt E, Souleau B, Nedellec G, Debuire B. Real-time quantitation of bcr-abl transcripts in haematological malignancies. Eur J Haematol. 2000 Oct;65(4):258-66. doi: 10.1034/j.1600-0609.2000.065004258.x. PMID 11073166
- [Background] Mitterbauer G, Nemeth P, Wacha S, Cross NC, Schwarzinger I, Jaeger U, Geissler K, Greinix HT, Kalhs P, Lechner K, Mannhalter C. Quantification of minimal residual disease in patients with BCR-ABL-positive acute lymphoblastic leukaemia using quantitative competitive polymerase chain reaction. Br J Haematol. 1999 Sep;106(3):634-43. doi: 10.1046/j.1365-2141.1999.01605.x. PMID 10468851
- [Background] Tabernero MD, Bortoluci AM, Alaejos I, Lopez-Berges MC, Rasillo A, Garcia-Sanz R, Garcia M, Sayagues JM, Gonzalez M, Mateo G, San Miguel JF, Orfao A. Adult precursor B-ALL with BCR/ABL gene rearrangements displays a unique immunophenotype based on the pattern of CD10, CD34, CD13 and CD38 expresssion. Leukemia. 2001 Mar;15(3):406-14. doi: 10.1038/sj.leu.2402060. PMID 11237064
- [Background] le Coutre P, Tassi E, Varella-Garcia M, Barni R, Mologni L, Cabrita G, Marchesi E, Supino R, Gambacorti-Passerini C. Induction of resistance to the Abelson inhibitor STI571 in human leukemic cells through gene amplification. Blood. 2000 Mar 1;95(5):1758-66. PMID 10688835
- [Background] Mahon FX, Deininger MW, Schultheis B, Chabrol J, Reiffers J, Goldman JM, Melo JV. Selection and characterization of BCR-ABL positive cell lines with differential sensitivity to the tyrosine kinase inhibitor STI571: diverse mechanisms of resistance. Blood. 2000 Aug 1;96(3):1070-9. PMID 10910924
- [Background] Weisberg E, Griffin JD. Mechanism of resistance to the ABL tyrosine kinase inhibitor STI571 in BCR/ABL-transformed hematopoietic cell lines. Blood. 2000 Jun 1;95(11):3498-505. PMID 10828035
- [Background] Gambacorti-Passerini C, Barni R, le Coutre P, Zucchetti M, Cabrita G, Cleris L, Rossi F, Gianazza E, Brueggen J, Cozens R, Pioltelli P, Pogliani E, Corneo G, Formelli F, D'Incalci M. Role of alpha1 acid glycoprotein in the in vivo resistance of human BCR-ABL(+) leukemic cells to the abl inhibitor STI571. J Natl Cancer Inst. 2000 Oct 18;92(20):1641-50. doi: 10.1093/jnci/92.20.1641. PMID 11036109
- See also: Spanish association of Haematology — http://www.aehh.org